CLINICAL TRIAL: NCT00421980
Title: An Open-Label, Multicentre, Long-Term Extension Study of Etanercept in Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-312
Record Dates: First submitted 2007-01-08; First posted 2007-01-15 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The primary objective of this study was to determine the long-term safety of etanercept in adults with AS who had completed study 0881A3-311-EU.

DETAILED DESCRIPTION:
This was an open-label, multicenter extension study that was conducted to evaluate the safety and efficacy of etanercept in the treatment of adult subjects with AS who had completed study 0881A3-311-EU. The study consisted of an open-label treatment period of up to approximately 96 weeks.

ELIGIBILITY:
1. Completed the entire 12 weeks of therapy in study 0881A3-311-EU, or completed at least 8 weeks of therapy and returned for the week 12 visit in study 0881A3-311-EU.
2. Negative serum β-HCG pregnancy test at baseline (all women of childbearing potential).
3. Sexually active women of childbearing potential had to use a medically acceptable form of contraception. Medically acceptable forms of contraception included oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception. Additionally, the use of condoms was suggested as an adjunct to the methods previously addressed to protect against sexually transmitted diseases and to provide additional protection against accidental pregnancy.
4. Sexually active men had to agree to use a medically accepted form of contraception during the study.
5. Able to reconstitute and self-inject test article or have a designee who can do so.
6. Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol-specific procedures were performed.
7. Able to store injectable test article at 2°C to 8°C.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2002-06; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Ghent, Belgium

REFERENCES:
- [Derived] Baraliakos X, Szumski AE, Kwok KK, Vlahos B, Borlenghi CE. Long-term Etanercept Response for Patients with Radiographic Axial Spondyloarthritis Based on Achievement of Early, Intermediate, or Late Responses During Index Studies. Rheumatol Ther. 2024 Jun;11(3):583-597. doi: 10.1007/s40744-024-00656-3. Epub 2024 Mar 15. PMID 38488976
- [Derived] Dijkmans B, Emery P, Hakala M, Leirisalo-Repo M, Mola EM, Paolozzi L, Salvarani C, Sanmarti R, Sibilia J, Sieper J, Van Den Bosch F, van der Heijde D, van der Linden S, Wajdula J. Etanercept in the longterm treatment of patients with ankylosing spondylitis. J Rheumatol. 2009 Jun;36(6):1256-64. doi: 10.3899/jrheum.081033. Epub 2009 May 1. PMID 19411393